CLINICAL TRIAL: NCT02619916
Title: Individual Mindfulness-Based Cognitive Therapy (MBCT) and Individual Cognitive Behavioral Therapy (CBT) for Depression in Patients After Cancer: a Randomized Controlled Trial
Brief Title: MBCT and CBT for Depression in Patients After Cancer: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other); Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Maya Schroevers, Dr. M. Schroevers, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-214
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Depressive Symptoms
Keywords: Cancer; Depression; MBCT; CBT
MeSH Terms: conditions — Depression; Neoplasms | interventions — Mindfulness-Based Cognitive Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MBCT (Experimental): Mindfulness-Based Cognitive Therapy
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (MBCT)
- CBT (Experimental): Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- TAU (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT) — The intervention consists of 8 weekly individual sessions of MBCT. Each session will be administered individually and will last 60 minutes
  Arms: MBCT
Behavioral: Cognitive Behavioral Therapy (CBT) — The intervention consists of 8 weekly individual sessions of CBT. Each session will be administered individually and will last 60 minutes.
  Arms: CBT

SUMMARY:
The purpose of this study is to determine whether mindfulness-based cognitive therapy (MBCT) and cognitive behavioral therapy (CBT) are effective in reducing depressive symptoms in patients after cancer

DETAILED DESCRIPTION:
Cancer patients are prone to develop depressive symptoms, even after curative treatment. Conventional therapies such as cognitive behavioral therapy (CBT) and mindfulness-based cognitive therapy (MBCT) are frequently used for reducing these depressive symptoms in patients with medical conditions. However, until now evidence from proper designed randomized controlled trials regarding the effectiveness of both interventions in cancer survivors, is lacking. Therefore, our longitudinal study aims to investigate the effectiveness of CBT and MBCT in reducing depressive symptoms in cancer survivors. In addition, potential moderators and mediators of each intervention will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Completion of curative cancer treatment (for primary diagnosis of cancer or possible recurrence of cancer) at least one year ago and no longer than five years ago.
* Currently no active cancer.
* ≥ 18 at the time of diagnosis of cancer and ≤ 75 at inclusion.
* Depressive symptoms as assessed by a Patient Health Questionnaire (PHQ-9) score ≥ 10 (indicating presence of at least mild depressive symptoms).
* Being able to read, write, and speak Dutch.

Exclusion Criteria:

* Severe psychiatric co-morbidity (i.e. acute suicidal ideations or behavior, recently experienced psychosis, diagnosis of schizophrenia, bipolar disorder, drug abuse or substance dependence, serious cognitive or neurological problems).
* Receiving psychological treatment for depressive symptoms, currently or less than two months prior to study participation.
* Unstable antidepressant medication regimen two months prior to inclusion of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in severity of depressive symptoms | pre-treatment (baseline) to post-treatment (approximately 3 months after baseline) and 3- and 9-month follow-up
  Severity of depressive symptoms will be assessed with the Beck Depression Inventory-II (BDI-II)

SECONDARY OUTCOMES:
Change in generalized anxiety | pre-treatment (baseline) to post-treatment (approximately 3 months after baseline) and 3- and 9-month follow-up
  Generalized anxiety is measured by the Generalised Anxiety Disorder Assessment (GAD 7)
Change in well-being | pre-treatment (baseline) to post-treatment (approximately 3 months after baseline) and 3- and 9-month follow-up
  Well-being is measured by the WHO Well-being Index (WHO-5)
Change in fear of recurrence | pre-treatment (baseline) to post-treatment (approximately 3 months after baseline) and 3- and 9-month follow-up
  Fear of recurrence will be measured by Concerns About Recurrence Scale (CARS)
Change in fatigue | pre-treatment (baseline) to post-treatment (approximately 3 months after baseline) and 3- and 9-month follow-up
  Fatigue is measured by the subsequent scale of the Multidimensional Fatigue Inventory (MFI-20)

CONTACTS AND LOCATIONS:
Overall Officials: Maya Schroevers, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Provincie Groningen, Netherlands